CLINICAL TRIAL: NCT07092956
Title: The Effect of Financial Literacy Education on Financial Literacy and Future Anxiety in Final Year Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Financial Literacy Education on Financial Literacy and Future Anxiety in Final-Year Nursing Students
Acronym: FLANURSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Miray Aksu, Assistant Professor of Nursing, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBU-HEM-MA-03; GATA-BAEK-2025/05-236 (Other: Gülhane Scientific Research Ethics Committee Approval No)
Record Dates: First submitted 2025-07-19; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Literacy; Anxiety and Fear; Nursing Students; Health Knowledge, Attitudes, Practice
Keywords: Financial Literacy; Future Anxiety; Nursing Students; Financial Education; Health Professions Education; Randomized Controlled Trial; Nurse Education
MeSH Terms: conditions — Literacy; Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model in which final-year nursing students were randomly allocated to either an experimental group receiving financial literacy training or a control group receiving no training. Pre- and post-tests were conducted for both groups to assess financial literacy and future anxiety. After post-intervention data collection, the control group was also provided with the same financial literacy education to ensure equal learning opportunity.
Masking Description: No masking was performed in this study. Both participants and investigators were aware of group assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Literacy Education (Experimental): Participants in this group received financial literacy education delivered by an expert in economics. The training covered budgeting, saving, investment tools, opportunity cost, and financial planning. Measurements were taken before and three weeks after the training.
  Interventions: Behavioral: Financial Literacy Education
- Control Group (No Intervention): Participants in this group did not receive any financial literacy education during the main study period. However, the same training was provided after post-intervention data collection to ensure ethical equity. Measurements were taken at the same intervals as in the experimental group.

INTERVENTIONS:
Behavioral: Financial Literacy Education — A structured financial literacy training program delivered by an expert in economics. The training includes topics such as budgeting, saving, opportunity cost, financial planning, and investment tools. It was provided to the experimental group over a single session, and outcomes were assessed three weeks later.
  Arms: Financial Literacy Education

SUMMARY:
This study aims to evaluate the effect of financial literacy education on financial literacy levels and future anxiety among senior-year nursing students. The research will be conducted at the University of Health Sciences, Gülhane Faculty of Nursing, using a randomized controlled trial design with pre-test and post-test measures. Participants will be selected from fourth-year nursing students enrolled in the 2024-2025 academic year. The intervention group will receive financial literacy training delivered by an expert in economics. The study will use the Financial Literacy Behavior and Attitude Scale and the Future Anxiety Scale for University Students to assess outcomes. The effectiveness of the training will be evaluated by comparing pre- and post-intervention data.

DETAILED DESCRIPTION:
his randomized controlled trial investigates the effectiveness of financial literacy education on improving financial literacy levels and reducing future anxiety among final-year nursing students. The intervention is designed to provide students with essential knowledge and skills related to budgeting, saving, opportunity cost, and financial planning, aiming to improve their confidence in managing personal finances and reducing anxiety about their future economic well-being.

Participants will be randomly assigned to either an experimental group receiving the educational intervention or a control group receiving no intervention during the main study period. Both groups will complete baseline (pre-test) and follow-up (post-test) assessments three weeks apart using the Financial Literacy Behavior and Attitude Scale and the Future Anxiety Scale for University Students. To ensure ethical equity, the control group will receive the same financial literacy education after the final assessments.

The study aims to provide evidence-based recommendations for incorporating financial literacy training into nursing curricula to better prepare students for their future professional and personal lives.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to voluntarily participate in the study
* Enrollment as a 4th-year nursing student at the University of Health Sciences, Gülhane Faculty of Nursing, during the 2024-2025 academic year
* No known hearing or visual impairments
* No prior participation in any financial literacy education

Currently employed in a paid part-time or full-time job

Exclusion Criteria:

* Voluntary withdrawal from the study at any point
* Incomplete participation in the study stages (e.g., missing pre-test or post-test data)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change in financial literacy scores | Baseline and 3 weeks post-intervention
  Financial literacy will be measured using the Financial Literacy Behavior and Attitude Scale (FODTÖ), which includes subdimensions such as spending, attitude, perception, and interest. Higher scores indicate greater financial literacy. As the score on the scale increases, future anxiety increases; as the score decreases, future anxiety decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Miray Aksu, Phd, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Gülhane Faculty of Nursing, Ankara, Etlik/Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No